CLINICAL TRIAL: NCT04290338
Title: Effects of the Premature Infant Oral Motor Intervention on the Oral Feeding Skills of the Premature Infants: A Randomized Controlled Trial
Brief Title: Effects of PIOMI on Oral Feeding of the Premature Infants
Acronym: PIOMI2020
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PIOMI2020Policlinico
Record Dates: First submitted 2020-02-24; First posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Feeding Disorder Neonatal

STUDY DESIGN:
Intervention Model Description: RCT characterized by the comparison between two groups (treated / untreated)
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PIOMI Group (Experimental): Patients in this group will receive the intraoral and extraoral stimulations provided by the PIOMI protocol. These stimulations will last 5 minutes and will be performed once a day for 7 consecutive days for each patient.
  Interventions: Other: PIOMI
- Control Group (No Intervention): Patients in this group will receive classic care.

INTERVENTIONS:
Other: PIOMI — Intraoral and extraoral stimulation.
  Arms: PIOMI Group

SUMMARY:
Randomized controlled clinical trial aimed at evaluating the effects of the "Premature infant oral motor intervention" method on the oral feeding skills of the premature infants.

DETAILED DESCRIPTION:
Numerous evidences emerge from the literature review on the usefulness of the PIOMI method to improve food skills in the premature infant. The goal of this study is to evaluate the effects of the PIOMI method by adding the gustatory stimulation to the original protocol.

ELIGIBILITY:
Inclusion Criteria:

* gestational age at birth between 25-33 weeks;
* clinical stability;
* possible presence of nasogastric or oro-gastric tube;
* non-invasive respiratory support (oxygen, high flows)

Exclusion Criteria:

* gestational age <25 weeks or> 33 weeks
* absence of clinical stability
* invasive respiratory support (CPAP)
* previous surgical interventions
* ongoing infections
* congenital and / or chromosomal diseases
* brain, metabolic, cardiac, gastrointestinal diseases
* presence of bronchopulmonary dysplasia

Ages: 25 Weeks to 33 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Mean volume | 7 days
  Mean volume of oral intake

SECONDARY OUTCOMES:
feeding efficiency | 3 days
  oral intake at day one and at day three
achievement of full oral feeding | 6 moths
  PMA on reaching full oral feeding
hospital stay time | 6 months
  days spending to the hospital
transition time | 6 months
  transition times from the tube to full oral feeding

CONTACTS AND LOCATIONS:
Overall Officials: Odoardo Picciolini, Study Director — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD may result in a publication.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 1 year